CLINICAL TRIAL: NCT05178641
Title: Overnight Pant Safety-in-use Diary Clinical Trial for Children With Nocturnal Enuresis
Brief Title: Overnight Pant Study for Children With Nocturnal Enuresis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: CSD2021096
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care (Experimental): For the first 3 weeks participants use Ninjamas Pyjama Pants, then for the next 3 weeks they switch to the Overnight Current Standard of Care.
  Interventions: Device: Ninjamas Pyjama Pants; Other: Participant's Overnight Current Standard of Care
- Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant (Experimental): For the first 3 weeks participants use their Overnight Current Standard of Care, then for the next 3 weeks they switch to Ninjamas Pyjama Pants.
  Interventions: Device: Ninjamas Pyjama Pants; Other: Participant's Overnight Current Standard of Care

INTERVENTIONS:
Device: Ninjamas Pyjama Pants — Disposable, absorbent underwear-like pyjama pant specifically designed to manage nocturnal enuresis in children by absorbing involuntary urine loss overnight and keeping the child's bed and clothing dry.
Other: Participant's Overnight Current Standard of Care — Any disposable or reusable absorbent diaper or pant product available on the US market that is used to absorb involuntary urine loss for children who are wetting the bed at night.

SUMMARY:
This study will evaluate the in-use tolerance of an absorbent disposable underwear pant developed for children with nocturnal enuresis by assessing adverse events. In addition product performance will be assessed by the parent at home via a daily diary.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for enrollment if the parent/legal guardian responds positively ("Yes") to the following questions:

1. Have you read, understood and signed the Informed Consent document?
2. Is your child generally healthy?
3. Is your child 4-7 years of age?
4. Does your child weigh approximately 37-63 pounds and fit into the test pant?
5. Thinking of the past 3 months, does your child wet the bed at night at least once per week?
6. Is your child currently using overnight pants or diapers?
7. Is your child willing to use their usual and/or supplied overnight pant products every night for the duration of the study?
8. Are you and your child willing to refrain from using wet wipes in the pant area for the duration of the clinical trial?
9. Are you willing to refrain from enrolling your child in other clinical or consumer studies for the duration of this clinical trial?
10. Are you and your child willing to refrain from using lotions, creams, ointments, oils, moisturizing bubble baths, powders, sunscreen and/or skin preparations in the child's pant area and on thighs for the duration of this clinical trial, unless required for medical reasons?
11. Are you and your child willing and able to comply with all study instructions?
12. Are you able to fill in the required questionnaires in English?

Exclusion Criteria:

Participants are ineligible for enrollment if the parent/legal guardian responds positively ("Yes") to any of the following questions:

1. Does your child have any acute or chronic skin conditions (excluding skin rash) in or around the pant area?
2. Does your child currently have (or have a history of) any significant illness or chronic medical condition?
3. Is your child currently using any medications?
4. Does your child currently wear absorbent products during the day?
5. Does your child suffer from any other lower urinary tract symptoms (e.g., increased frequency, daytime incontinence, urgency, genital, or lower urinary tract pain) or a history of bladder dysfunction?

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Huesing-Wray, Principal Investigator — North Cliff Consultants
Locations (1):
- North Cliff Consultants, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment and enrollment was done by a Clinical Research site, North Cliff Consultants, Inc. in the Cincinnati, Ohio area.
Pre-assignment Details: Participants were given 4 days practice time to get used to the study procedures (Jan 13th - Jan 16th), before the first period started on Jan 17th.
Period: First 3 Weeks of Study (Week 1-3)
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant
Started | 16 | 16
Completed | 12 | 14
Not Completed | 4 | 2
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Last 3 Weeks of Study (Week 3-6)
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant
Started | 12 | 14
Completed | 12 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 16 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 9 | 14 | 23
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Height [Mean (Full Range); unit: Inches] | 44.5 [42 to 48] | 45.1 [40 to 51] | 44.8 [40 to 51]
Weight [Mean (Full Range); unit: LBS] | 44.9 [37.4 to 56] | 45.0 [34 to 61.6] | 45.0 [34 to 61.6]
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin type is a numerical classification schema for human skin color ranging from I (fair skin) to IV (dark skin).
  Participants
    Fitzpatrick I | 0 | 0 | 0
    Fitzpatrick II | 1 | 5 | 6
    Fitzpatrick III | 7 | 7 | 14
    Fitzpatrick IV | 5 | 2 | 7
    Fitzpatrick V | 3 | 1 | 4
    Fitzpatrick VI | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number, Frequency and Severity of Product Related Adverse Events
Description: Adverse Device Effect and Adverse Event tracking twice daily via a safety in-use diary.
Time Frame: From admission to discharge, up to 6 weeks
Measure: Number; unit: Number of product related Adverse Events
Groups:
- Total: All participants who participated in the study
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant | Total
Number analyzed (Participants) | 16 | 16 | 32
Number of product related Adverse Events
  Diaper Dermatitis | 47 | 63 | 110
  Pruritus in diaper area | 5 | 4 | 9
  Feeling of heat in crotch area | 1 | 2 | 3
  Serious Adverse Events | 0 | 0 | 0
  Product related Adverse Events with causality assessed by PI as doubtful | 47 | 63 | 110

2. Secondary Outcome: Parent Assessed Product Performance in Terms of Urine Leaking
Description: Daily urine leakage diary (yes/no) reported every morning by parent via visual inspection of presence of wet stain on bed sheet and location of wet stain on clothes. Only participants who completed both periods and had at least one overnight pant per period with a urine load were included in this analysis. An overnight pant was considered urine loaded when the overall pant weight exceeded 1.1 ounce (oz). The number of leaks for each treatment option was calculated as number of leakage observations answered with "yes".
Time Frame: From admission to discharge, up to 6 weeks
Population: Only participants who completed both periods and had at least one overnight pant per period with a urine load were included in this analysis. An overnight pant was considered loaded when the overall pant weight exceeded 1.1 ounce (oz).
Measure: Number; unit: Number of pants with reported leaks
Units Other Than Participants: Number of pants with a urine load
Groups:
- Total: All participants in the study who completed both periods
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant | Total
Number analyzed (Participants) | 12 | 14 | 26
Number analyzed (Number of pants with a urine load) | 369 | 395 | 764
Number of pants with reported leaks
  Treatment Effect of Ninjamas Pyjama Pant: number analyzed (Number of pants with a urine load) | 196 | 196 | 392
  Treatment Effect of Ninjamas Pyjama Pant | 2 | 0 | 2
  Treatment Effect of Participant's Overnight Current Standard of Care: number analyzed (Participants) | 11 | 14 | 25
  Treatment Effect of Participant's Overnight Current Standard of Care: number analyzed (Number of pants with a urine load) | 173 | 199 | 377
  Treatment Effect of Participant's Overnight Current Standard of Care | 8 | 3 | 11
  Treatment effect of both periods combined | 10 | 3 | 13

ADVERSE EVENTS:
Time Frame: 6 weeks (Jan 13th - Feb 28, 2022)
Groups:
- Ninjamas Pyjama Pant: For either the first 3 weeks of the study or the last 3 weeks of the study participants used Ninjamas Pyjama Pants, depending on randomization.
  Ninjamas Pyjama Pants: Disposable, absorbent underwear-like pyjama pant specifically designed to manage nocturnal enuresis in children by absorbing involuntary urine loss overnight and keeping the child's bed and clothing dry.
- Participant's Overnight Current Standard of Care: For either the first 3 weeks of the study or the last 3 weeks of the study participants used their Overnight Current Standard of Care.
  Participant's Overnight Current Standard of Care: Any disposable or reusable absorbent diaper or pant product available on the US market that is used to absorb involuntary urine loss for children who are wetting the bed at night.
Arm/Group | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant | Ninjamas Pyjama Pant | Participant's Overnight Current Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 12/16 | 14/16 | 21/30 | 19/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ninjamas Pyjama Pant, Then Participant's Overnight Current Standard of Care (N=16) | Participant's Overnight Current Standard of Care, Then Ninjamas Pyjama Pant (N=16) | Ninjamas Pyjama Pant (N=30) | Participant's Overnight Current Standard of Care (N=28)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 11 | 11 | 17 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 4 | 6 | 6 — Localized itching in diaper area
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 2
Ear Infection (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Covid-19 (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Tooth Abscess (Infections and infestations) | 0 | 1 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Feeling hot (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 — Sensation of heat in crotch area
Pyrexia (General disorders) | 1 | 1 | 1 | 1 — Fever
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 — Allergy with cold symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT05178641/Prot_SAP_000.pdf